CLINICAL TRIAL: NCT07033728
Title: The Health of Women Monitored in the Addiction Department of the Strasbourg University Hospitals
Acronym: Santé-Fem
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9616
Record Dates: First submitted 2025-05-16; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-05

CONDITIONS: Drug Addiction
Keywords: Drug Addiction; Addiction
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The health of women suffering from addiction is little known and little explored in the literature. Indeed, they represent only 20% of addicted patients in general and are encountered primarily during pregnancy or complex situations involving young children.

In the Addiction Department of Strasbourg University Hospitals, the investigators have established a midwifery consultation exclusively for women of all ages.

During the treatment of the women, the investigators were able to identify the specific issues faced by women suffering from addiction and the specific care requirements for this population.

ELIGIBILITY:
Inclusion Criteria:

* Female, adult (≥ 18 years old)
* Undergoing follow-up at the CSAPA Addictions Department of the HUS
* Having met the team's midwife at least once
* Absence of written objection in the patient's medical record regarding the reuse of her data for scientific research purposes.

Exclusion Criteria:

* Absence of written objection in the patient's medical record regarding the reuse of her data for scientific research purposes
* Female minor
* Female who has not initiated follow-up with the CSAPA team
* Women who have never had a consultation with the team's midwife

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female, adult (≥ 18 years old) undergoing follow-up at the CSAPA Addictions Department of the HUS
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2026-09-24 (Estimated); Study Completion 2026-09-24 (Estimated)

PRIMARY OUTCOMES:
Rate of gynecological follow-up regardless of age compared to the general population | Up to 18 months
  This is a retrospective study to carry out an inventory of the health status of women treated at the CSAPA (Center for Addiction Care, Support, and Prevention) of the HUS (University Hospitals of Strasbourg)

SECONDARY OUTCOMES:
Rate of Consumption of toxic drugs compared to the general population | Up to 18 months
  This is a retrospective study to carry out an inventory of the health status of women treated at the CSAPA (Center for Addiction Care, Support, and Prevention) of the HUS (University Hospitals of Strasbourg)
Rate of sexual violence compared to the general population | Up to 18 months
  This is a retrospective study to carry out an inventory of the health status of women treated at the CSAPA (Center for Addiction Care, Support, and Prevention) of the HUS (University Hospitals of Strasbourg)

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'addictologie - CHU de Strasbourg - France, Strasbourg, France